CLINICAL TRIAL: NCT03376464
Title: Prospective Evaluation of Xeomin Cosmetic in the Management of the Masseter Using Two Different Injection Techniques
Brief Title: Xeomin Cosmetic in the Management of Masseter
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-01-001
Record Dates: First submitted 2017-12-10; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Masseter Muscle Hypertrophy
Keywords: Xeomin Cosmetic;; Masseteric Hypertrophy
MeSH Terms: conditions — Masticatory Muscles, Hypertrophy of

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single injection technique (SIT) (Experimental): 40 U of Xeomin Cosmetic delivered directly into the region where the three masseter heads overlap.
  Interventions: Device: Xeomin Cosmetic
- multi-injection technique (MIT) (Experimental): A distribution of 40 U (8 U distributed in 5 different areas) of Xeomin Cosmetic over the width of the masseter while respecting the upper limit of the anterior border of the masseter and the inferior insertion of the masseter. The injections are separated by a 1cm distance and the dose is equally distributed across these sites.
  Interventions: Device: Xeomin Cosmetic

INTERVENTIONS:
Device: Xeomin Cosmetic — Xeomin Cosmetic is the purest commercially available botulinum toxin type A available to date. It has been approved by Health Canada since 2012 for the temporary improvement in the appearance of moderate to severe glabellar lines.

SUMMARY:
The goal of this study was to evaluate the efficacy and safety of two injection techniques in the management of masseteric hypertrophy using Xeomin Cosmetic.

DETAILED DESCRIPTION:
Background: Xeomin Cosmetic has been used previously in the management of masseteric hypertrophy. However, a standardized injection technique has not been established. The goal of the present study was to evaluate the efficacy and safety of two injection techniques in the management of masseteric hypertrophy using Xeomin Cosmetic.

Methods: Thirty female patients with masseteric hypertrophy were recruited and evenly randomized to receive bilateral treatments of either 1) a single injection technique (SIT), or 2) a multi-injection technique (MIT). Improvement of masseteric hypertrophy was assessed at Week 16 using standardized measurements and photographs. Patients completed a 5-point satisfaction questionnaire while physicians the global aesthetic improvement scale (GAIS) and 10-point photonumeric masseter prominence rating scale.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of consent, women over the age of 18 years old.
2. Patients with established hypertrophy of the masseters, palpable and visible.
3. Accepted the obligation not to receive any other facial procedures through the 6-month follow-up.
4. Understood and accepted the obligation and would be logistically able to appear for all scheduled follow-up visits.
5. No previous facial fillers for a period of 6 months prior to this study.
6. No previous facial fillers along the jawline for 18 months
7. Capable of providing informed consent.
8. No previous botulinum toxin type A treatment for masseteric hypertrophy in the last 12 months.

Exclusion Criteria:

1. Current Pregnancy or lactation
2. Hypersensitivity to Xeomin
3. Generalized disorders of muscle activity (e.g. myasthenia gravis, Lambert Eaton syndrome)
4. Presence of infection at the site of injection
5. Inability to comply with follow-up and abstain from facial injections during the study period
6. Patients with a score of 2 or greater on the Merz Aesthetics Scale for the Jawline

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Metric masseteric hypertrophy improvement outcomes between SIT and MIT at 16 weeks in comparison to baseline. | Baseline to 16 weeks
  The difference in physician assessed efficacy using standardized masseter improvement measurements between two different injection techniques at 16 weeks (visit 4) in comparison to baseline (visit 2).

SECONDARY OUTCOMES:
Masseter photo-numeric aesthetic rating scales between SIT and MIT at 16 weeks in comparison to baseline. | Baseline to 16 weeks
  Face shape and masseteric prominence rating
Patient Satisfaction Questionnaire | Baseline to 20 weeks
Global Aesthetic Improvement Scale | Baseline to 20 weeks

OTHER OUTCOMES:
Adverse Events | Baseline to 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, MD, Principal Investigator — Erevna Innovations Inc.

IPD SHARING:
Plan to Share IPD: No